CLINICAL TRIAL: NCT06282705
Title: Is There a Dose-response Effect on Bone Characteristics in Relation to Drop Jump Height?
Brief Title: Dose Response Effect of Drop Jumps on Bone Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, Ian Varley, Associate Professor, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 306347
Record Dates: First submitted 2024-02-07; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy Participants; Low Activity Level
Keywords: Bone; Osteogenic activity; External Load; Drop jumps

STUDY DESIGN:
Intervention Model Description: Semi-randomised, matched model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 cm Diagonal drop jump (Experimental): Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 0 cm (floor). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Interventions: Behavioral: Diagonal Drop Jumps 0cm
- 40 cm diagonal drop jump (Experimental): Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 40 cm (plyometric box). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Interventions: Behavioral: Diagonal Drop Jumps 40cm
- 60 cm diagonal drop jump (Experimental): Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 60 cm (plyometric box). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Interventions: Behavioral: Diagonal Drop Jumps 60cm
- Control (No Intervention): No exercise intervention performed.

INTERVENTIONS:
Behavioral: Diagonal Drop Jumps 0cm — Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 0 cm (floor). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Arms: 0 cm Diagonal drop jump
Behavioral: Diagonal Drop Jumps 40cm — Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 40 cm (plyo box). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Arms: 40 cm diagonal drop jump
Behavioral: Diagonal Drop Jumps 60cm — Participants will complete 4 unsupervised home drop jump sessions per week ( minimum 24 hours between each session) for the duration of the study (e.g., Mon, Wed, Fri, Sun) from a height of 60 cm (plyo box). They will perform 20 diagonal drop jumps on each side (20 x dropping left and 20 x dropping right) with 30 seconds between each jump. The routine will be demonstrated in full on the first laboratory session. The intervention will last 16 weeks.
  Arms: 60 cm diagonal drop jump

SUMMARY:
The study aims to assess if a 16-week drop jump intervention from different heights shows different bone adaptations. Participants will complete four visits over a period of 16 weeks. An initial consultation will be conducted to ensure participants meet the inclusion criteria following participant recruitment. Estimated load being applied to the bone, will be assessed using non-invasive biomechanical procedures (Inertial Measurement Units, motion analysis, force plates) during drop jumps. Participants will be assigned a drop jump height of 0 cm, 30 cm or 60 cm based on a significant difference in external load at these heights or assigned to a control group where no jumps will be performed. Groups will be matched for body mass to ensure that jump height produces the load. The participants will be asked to perform 40 jumps (20 each side), 4 times per week ensuring jumping bouts are separated by 24 hours. Bone characteristics will be assessed via whole body dual-energy X-ray absorptiometry (DXA) scans and bilateral peripheral Quantitative Computed Tomography (pQCT) scans. Lab based jumping will take place on week 0, week 6, week 12, and week 16 to understand the loading applied during the different jump height groups. pQCT scans will take place on week 0, week 12, week 16 and DXA scans will take place week 0 and week 16. The reasoning of week 12 for pQCT being it may show a significant timepoint for bone formation during the remodelling cycle. During visits participants will complete a health screen, the Bone specific Physical Activity Questionnaire (BPAQ), a food frequency questionnaire and Pittsburgh sleep quality questionnaire alongside consent as tools to monitor any changes to participant lifestyle across the study. Differences in bone characteristics, lab measures and jump heights will be analysed between and within participants.

The present study aims to use varied drop jump heights to identify an osteogenic dose response effect. Drop jumps have been previously used to expose osteogenic effects in research due to the load produced at impact. Is it possible to identify an optimum height for bone response during impact? If so do we then find anything above this height actually has negative or no effect on a group of individuals?

DETAILED DESCRIPTION:
There are few studies that attempt to identify optimal exercises for bone health with specific loading variables being quantified. The identification of an osteogenic threshold during single or multiple activity bouts would allow us to understand the optimal volume/magnitude of exercise/loading that causes an osteogenic response. Understanding the optimal exercise characteristics for osteogenesis will subsequently allow specific bone enhancing exercise to be prescribed. Currently, ambiguity exists as in the guidance for optimising bone health through exercise, for example, a recently published position statement on increasing peak bone mass in adolescents recommends that 5-6 months of vigorous physical activity should be performed but does not quantify the specific speed or intensity of activity required.

pQCT and DXA will be used to measure bone characteristics. Both methods are a common way of obtaining data detailing bone architecture and geometry within established research establishments including universities and National Health Service (NHS) trusts. Through pQCT, bone geometry, both cortical and trabecular bone can be measured and as a result, bone quality can be assessed. Bone measurement via pQCT is widely used in research and is a non-invasive method of imaging bone to provide estimates of bone strength in the peripheral skeleton to differentiate cortical from trabecular bone and assess bone geometry and density. DXA is the gold standard method of measuring bone mineral density and is commonly used to assess osteoporosis risk.

In addition, body composition (which will be derived from the DXA) may be associated with bone characteristics due to body mass and composition relating to bone loading and muscle acting on bone to produce bone strain.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 years old
* Have a low physical activity status defined as partaking in physical training activities no more than 2x per week.
* No current regular participation (more than once per week) in exercise programmes known to influence bone inc. gymnastics, dance, court sports, ball sports or racquet sports.
* Be able to travel to the laboratory using a vehicle or public transport
* Have the ability to comprehend and understand communication and instruction in English in order to consent and safely participate in study.
* Have no current unresolved cardiovascular complaints to avoid any cardiovascular complications when performing activities of daily living.

Exclusion Criteria:

* Prescribed medication that influences bone metabolism such as corticosteroids, anticancer drugs, and diabetes related Drugs
* Joint replacement or prostheses
* Currently or recently injured
* Medical conditions adversely affected by exposure to ionising radiation.
* History of high levels of ionising radiation exposure (e.g., medical treatment).
* Breastfeeding women, pregnant women and women trying to become pregnant
* Females who are on any form of contraception that may influence changes in bone
* Females who have current or previous history of an endocrine disorder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
BMD as assessed by whole body dual-energy X-ray absorptiometry (DXA). | From baseline (week 0) to end of intervention (week 16)
  Bone mineral density (BMD)
BMC as assessed by whole body dual-energy X-ray absorptiometry (DXA). | From baseline (week 0) to end of intervention (week 16)
  Bone mineral content (BMC)
Total bone area as assessed by whole body dual-energy X-ray absorptiometry (DXA). | From baseline (week 0) to end of intervention (week 16)
  Total bone area
Trabecular density as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  Trabecular density measured at the 4% site of the tibia length.
Cortical thickness as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  Cortical thickness measured at the 14% and 38% site of the tibial length.
Periosteal circumference as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  Periosteal circumference measured at the 14% and 38% site of the tibial length.
Axial bone strength (SSIX) as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  SSIX measured at the 14% and 38% site of the tibial length.
Axial bone strength (SSIY) as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  SSIY measured at the 14% and 38% site of the tibial length.
Polar bone strength (SSIPOL) as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  SSIPOL measured at the 14% and 38% site of the tibial length.
Cortical density as assessed by peripheral quantitative tomography (pQCT) of tibia. | From baseline (week 0) to mid intervention (week 12) and end of intervention (week 16)
  Cortical density measured at the 14%, 38% and 66% site of the tibial length.

SECONDARY OUTCOMES:
Peak impact load as assessed by force plates. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Peak impact load derived from ground reaction force (GRF)
Impulse as assessed by force plates. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Impulse derived from ground reaction force (GRF)
Load rate as assessed by force plates. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Load rate derived from ground reaction force (GRF)
Jump height as assessed by force plates. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Jump height derived from ground reaction force (GRF)
Centre of Mass (CoM) velocity as assessed by force plates. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  CoM velocity derived from ground reaction force (GRF)
Peak acceleration as assessed by Inertial measurement units (IMU). | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Peak accelerations calculated from tibial mounted IMUs.
Stiffness as assessed by motion capture. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Knee and ankle Stiffness derived from motion capture.
Moments as assessed by motion capture. | From baseline (week 0) to mid intervention (week 6, week 12) and end of intervention (week 16)
  Knee and ankle moments derived from motion capture.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kenkre JS, Bassett J. The bone remodelling cycle. Ann Clin Biochem. 2018 May;55(3):308-327. doi: 10.1177/0004563218759371. Epub 2018 Mar 4. PMID 29368538
- [Background] Min SK, Oh T, Kim SH, Cho J, Chung HY, Park DH, Kim CS. Position Statement: Exercise Guidelines to Increase Peak Bone Mass in Adolescents. J Bone Metab. 2019 Nov;26(4):225-239. doi: 10.11005/jbm.2019.26.4.225. Epub 2019 Nov 30. PMID 31832388